CLINICAL TRIAL: NCT01444170
Title: A Single Site Double Blind Placebo Controlled Study of the Effects of a Dietary Supplement on Muscle Recovery Following Exercise-Induced Muscle Damage
Brief Title: Nutritional Supplement, Eccentric Exercise and Recovery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Iovate Health Sciences International Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-316-2006; UPN06050404
Record Dates: First submitted 2008-01-30; First posted 2011-09-30 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Injury; Inflammation
Keywords: eccentric exercise; exercise induce muscle damage; isometric strength; range of motion; self report symptoms; mechanical pain threshold
MeSH Terms: conditions — Wounds and Injuries; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sugar pill (Placebo Comparator): Placebo "sugar" pill was used as a sham control
  Interventions: Drug: placebo sugar pill
- dicreatinol sulfate (Experimental)
  Interventions: Dietary Supplement: dicreatinol sulfate; Drug: placebo sugar pill

INTERVENTIONS:
Dietary Supplement: dicreatinol sulfate — nutritional supplement
  Other Names: Sham control
  Arms: dicreatinol sulfate
Drug: placebo sugar pill

SUMMARY:
The objectives of this study are to assess the effectiveness of a nutritional supplement on muscle functional recovery following induced muscle damage from high intensity resistance exercise. The investigators hypothesize that a short-term dietary supplementation will significantly improve muscle functional recovery following an intense bout of eccentric exercise compared to a placebo.

DETAILED DESCRIPTION:
Impaired or incomplete recovery following high intensity exercise can negatively affect physical performance and delay functional progression, thereby reducing an athlete's chance of performing at his or her peak level. Athletes are constantly seeking ways to speed muscle recovery from strenuous exercise and muscle damage. Anabolic steroids are potent stimulators of muscle growth and repair and have been used extensively by athletes to hasten structural and functional recovery during peak periods of strenuous training. However, anabolic steroids are classified as banned substances by all major sports organizing committees that oversee and regulate amateur and professional athletics. In addition long-term use of anabolic steroids has known side effects that can negatively impact an athlete's health status. Dietary supplements are safe and viable alternatives that, if taken in the optimal doses, can provide positive effects on muscle growth and repair and ultimately human performance. Athletes have used dietary supplements extensively to facilitate tissue growth and repair following muscle-damaging events such as high-intensity resistance exercise and participation in contact sports. Following intense resistance exercise, an acute inflammatory response drives the repair process by synthesizing and releasing chemical mediators locally in the injured muscle. Inflammatory mediators help attract growth factors used for protein synthesis. The inflammatory response has also been shown to produce high levels of oxygen-derived free radicals that if allowed to proceed unabated, can produce further muscle damage, thus hindering the repair process. A protein-based dietary supplement, if taken in the optimal dosing schedule, may enhance the recovery process by blunting the magnitude of the acute inflammatory response and facilitating growth and repair through increased protein synthesis in damaged muscle tissue. Understanding the nutritional requirements of athletes engaged in high intensity training and competition is necessary to insure adequate recovery between exercise bouts. This will improve training and functional gains as well as act as a prophylaxis to skeletal muscle injury.

The objectives of this study are to assess the effectiveness of a nutritional supplement on muscle functional recovery following induced muscle damage from high intensity resistance exercise. This will be accomplished by evaluating baseline changes over the course of the recovery phase on severity of the symptomatic response and functional impairment in post-exercise skeletal muscle damage. The biceps brachii muscle will be targeted for this study. The investigators have established a safe and effective experimental arm curl model for inducing skeletal muscle soreness and dysfunction in human subjects using eccentric exercise to the bicep brachii muscle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smoking
* Untrained young adult males and females (age 18-25 years)
* Free of vitamin/mineral supplementation for six weeks prior to the study

Exclusion Criteria:

* Pregnant or positive pregnancy test
* Persons involved in a regular weight-training program within the last six weeks or with a prior history (within the last 6 weeks) of injury to the biceps brachii or elbow region
* Recent history or current reported use of anti-inflammatory medication, and active weight loss > 5 kg in prior 3 months (intended or unintended)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2006-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in self-reported symptoms and functional impairment at 10 days, 12 days, 14 days, 17 days and 20 days | 20 days

SECONDARY OUTCOMES:
Change from baseline in elbow range-of-motion at 10 days, 12 days, 14 days, 17 days and 20 days | 20 days
Change from baseline in biceps brachii isometric strength at 10 days, 12 days, 14 days, 17 days and 20 days | 20 days
Change from baseline in Mechanical Pain Threshold at 10 days, 12 days, 14 days, 17 days and 20 days | 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Borsa, PhD, Principal Investigator — University of Florida
Locations (1):
- Center for Exercise Science, Gainesville, Florida, United States

REFERENCES:
- See also: Iovate Health Sciences Research, Inc. — http://www.iovate.com